CLINICAL TRIAL: NCT07364240
Title: The Effect of Person-Centered Occupational Therapy Interventions on Occupational Performance, Self-Efficacy and Psychological Resilience in Substance Use Disorder
Brief Title: Effect of Person-Centered Occupational Therapy Interventions for Substance Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Büşra Yuvalı, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-215
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Substance Use Disorder (SUD)
Keywords: occupational therapy; Person- centered intervention; Occupational Performance; Self Efficacy; Psychological Resilience
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Participants in this group will receive person-centered occupational therapy interventions in addition to their routine treatment.
  Interventions: Behavioral: Person-Centered Occupational Therapy
- Control Group (Active Comparator): Participants in this group will receive a one-time awareness training session about substance use disorder and its effects, in addition to their routine clinical follow-up.
  Interventions: Behavioral: Awareness Training

INTERVENTIONS:
Behavioral: Awareness Training — A single-session educational program designed to increase awareness about the consequences of substance use and the recovery process.
  Arms: Control Group
Behavioral: Person-Centered Occupational Therapy — An 8-week person-centered program (3 sessions per week) focusing on daily life activities, productivity, and leisure goals identified through the COPM.
  Arms: Study Group

SUMMARY:
This study investigates the impact of person-centered occupational therapy interventions on individuals diagnosed with substance use disorder. Substance use often leads to isolation and difficulties in daily activities such as work, self-care, and leisure time. The research aims to evaluate how a tailored 8-week therapy program affects participants' occupational performance, self-efficacy, and psychological resilience. Participants will be divided into a study group receiving therapy and a control group.

DETAILED DESCRIPTION:
Participants aged 18-65 with a DSM-5 diagnosis of substance use disorder will be recruited from the Erenköy AMATEM unit. The study employs an experimental design with 34 participants (17 in the study group, 17 in the control group). The study group will receive person-centered occupational therapy interventions 3 times per week for a total of 8 weeks.

The intervention process is based on the four stages of person-centered practice: identifying occupational performance problems using the Canadian Occupational Performance Measure (COPM), brainstorming realistic goals, implementing tailored strategies (e.g., time management, vocational skills, or healthy habits), and revising the process based on feedback . Assessment tools including the COPM, Self-Efficacy Scale, and Brief Resilience Scale will be administered at baseline and after the 8-week intervention to measure changes in performance and psychological factors.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with substance use disorder according to DSM-5 criteria.
* Having completed the detoxification process.
* Being between the ages of 18-65.
* Having at least a primary school education.
* Volunteering to participate and signing the informed consent.

Exclusion Criteria:

* Being in an acute psychotic episode.
* Having severe neurological deficits that prevent responding to assessments. -Having severe visual or hearing loss that prevents completing the test batteries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | Change from baseline at 8 weeks.
  A semi-structured interview used to identify and prioritize everyday activities that the individual finds difficult to perform. It measures two components: Occupational Performance and Satisfaction. Both are scored on a scale of 1 to 10, where higher scores indicate better performance and higher satisfaction.

SECONDARY OUTCOMES:
Self-Efficacy Scale | Change from baseline at 8 weeks.
  A 23-item scale measuring the individual's self-judgment of their ability to achieve intended goals. Scores range from 23 to 115, with higher scores indicating higher self-efficacy.
Brief Resilience Scale | Change from baseline at 8 weeks
  A 6-item self-report scale measuring the individual's ability to bounce back or recover from stress. Higher scores indicate higher psychological resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Onur Altuntaş, Assoc Prof, Study Director — Hacettepe University; Büşra Yuvalı, PhD Cand, Principal Investigator — Hacettepe University
Locations (1):
- Erenköy Mental and Neurological Diseases Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No